CLINICAL TRIAL: NCT03012269
Title: The Study on the Brain Mechanisms for the Rehabilitation of Working Memory Deficits in Patients With Acquired Brain Injury Using Multimodal Magnetic Resonance Imaging
Brief Title: The Neural Substrates for Working Memory Training
Acronym: WMT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Rehabilitation Research Center (Other Government)
Responsible Party: Principal Investigator, Yun XiaoPing, Director of Department of Rehabilitation Evaluation, China Rehabilitation Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSFC-81272165
Record Dates: First submitted 2016-12-31; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Rehabilitation; Working Memory

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Working Memory Training (Experimental): The subjects of experimental group received a series of working memory training, 30 min for 5 days per week during 6 weeks.
  Interventions: Behavioral: Working memory training
- Non-Working Memory Training (No Intervention): The subjects of control group performed traditional cognitive rehabilitation without working memory training, 30 min for 5 days per week during 6 weeks.

INTERVENTIONS:
Behavioral: Working memory training
  Arms: Working Memory Training

SUMMARY:
This study aims to conduct a contrast study on the characteristics of functional and structural connectivity of neural networks of working memory in patients with acquired brain injury versus normal controls, using resting-state functional connectivity magnetic resonance imaging, task-specific functional magnetic resonance imaging and diffusion tensor imaging, combined with cognitive behavioral examinations. Another purpose is to reveal the characteristics of dynamic change of neural networks of working memory pre- and post-intervention in patients with working memory dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Right handedness
* Diagnosis of traumatic brain injury or stroke
* Course of disease within one year
* The score of MoCA test > 24
* Able to understand instructions

Exclusion Criteria:

* Aphasia, unilateral spatial neglect, agnosia, apraxia
* Hearing impairment or visual impairment
* History of taking psychiatric drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-10; Primary Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Training-induced brain activations during working memory tasks in fMRI | six weeks
  Training-induced increased and decreased brain activations (Number of voxels) during n-back verbal WM task compared to the pre-training baseline

SECONDARY OUTCOMES:
The fluid intelligence measured by Raven's Standard Progressive Matrices (RSPM) test | six weeks
Attention ability assessed by Stroop color-word test | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Yun, MD, Principal Investigator — Department of Rehabilitation Evaluation, China Rehabilitation Research Center
Locations (1):
- Department of Rehabilitation Evaluation, China Rehabilitation Research Center, Beijing, Beijing Municipality, China